CLINICAL TRIAL: NCT01859494
Title: Performance of the Ninja 3 Blood Glucose Monitoring System
Brief Title: Evaluation of an Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2012-009-01
Record Dates: First submitted 2013-05-19; First posted 2013-05-22 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Users of the Monitoring System (Experimental): Untrained subjects with diabetes used the NINJA 3 Investigational Blood Glucose Monitoring System.
  Interventions: Device: NINJA 3 Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: NINJA 3 Investigational Blood Glucose Monitoring System — Untrained subjects with diabetes self-tested capillary fingerstick and palm blood using the NINJA 3 Investigational Blood Glucose Monitoring System. Study staff tested subject fingerstick blood. All BG results were compared to reference method results obtained from subject capillary plasma.

SUMMARY:
The purpose of this study was to determine if untrained subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 years of age and older
2. People with type 1 or type 2 diabetes
3. Able to speak, read, and understand English
4. Willing to complete all study procedures

Exclusion Criteria:

1. Hemophilia or any other bleeding disorder
2. Pregnancy
3. Physical, visual, or neurological impairments that would make the person unable to perform testing with the BGM
4. Previously participated in a BG monitor study using the Ninja 3 BGMS
5. Working for a medical laboratory, hospital, or other clinical setting that involves training on and clinical use of blood glucose monitors
6. Working for a competitive medical device company, or having an immediate family member who works for such a company
7. A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk.

The enrollment criteria for the study population:

1. At least 60% of subjects will be younger than age 65
2. At least 20% of subjects will have type 1 diabetes
3. At least 50% of subjects with type 2 diabetes wil be insulin users.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute; Leslie J Klaff, MD, Principal Investigator — Rainier Clinical Research Center
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
When it is cleared, results data will be provided.

RESULTS

PARTICIPANT FLOW:
Groups:
- Users of the Monitoring System: Untrained subjects with diabetes used the NINJA 3 Investigational Blood Glucose Monitoring System.
  NINJA 3 Investigational Blood Glucose Monitoring System: Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the NINJA 3 Investigational Blood Glucose Monitoring System. Study staff tested subject fingerstick blood. All BG results were compared to reference method results obtained from subject capillary plasma.
Period: Overall Study
Arm/Group | Users of the Monitoring System
Started | 219
Completed | 218
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Two subjects were screen failures due to not meeting enrollment criteria. 221 consented but only 219 enrolled into study.
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 221
Age, Continuous [Mean (Full Range); unit: years] | 51.8 [18 to 95]
Gender [Count of Participants; unit: Participants]
  Female | 108
  Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 197
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Number; unit: participants] — Subjects provided more than one choice for Race, therefore the apparent frequency total for Race was different from the number of subjects.
  participants
    American Indian or Alaska Native | 4
    Asian | 9
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 10
    White | 194
    More than one race | 3
    Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 221

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/-15mg/dL (<75mg/dL) or Within +/-20% (>=75mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 218 (219-1) Blood glucose results were analyzed. One subject discontinued from testing after low Blood Glucose (BG) fingerstick result (hypoglycemia AE), thus no reference result available for that subject.
Measure: Number; unit: Blood Glucose results within 15mg/dL/20%
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 218
Blood Glucose results within 15mg/dL/20% | 218

2. Secondary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG)Results Within +/- 15mg/dL (<100mg/L YSI) or Within +/- 15% (>=100mg/dL YSI) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI BG results were used to calculate the number of BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) or +/- 15% (>=100mg/dL YSI capillary plasma)
Time Frame: 1 hour
Population: 218 (219-1) Blood glucose results were analyzed. One subject discontinued from testing after low BG fingerstick result (hypoglycemia AE), thus no reference result available for that subject.
Measure: Number; unit: Blood Glucose results within 15mg/dL/15%
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 218
Blood Glucose results within 15mg/dL/15% | 215

3. Secondary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG)Results Within +/- 12.5mg/dL (<100mg/L YSI) or Within +/- 12.5% (>=100mg/dL YSI) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI BG results were used to calculate the number of BGMS results within +/- 12.5mg/dL (<100mg/dL YSI capillary plasma) or +/- 12.5% (>=100mg/dL YSI capillary plasma)
Time Frame: 1 hour
Population: as for outcome 2
Measure: Number; unit: Bld Glucose results w/in 12.5mg/dL/12.5%
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 218
Bld Glucose results w/in 12.5mg/dL/12.5% | 214

4. Secondary Outcome: Number of Glucose Results From Alternative Site Testing (AST) of the Palm Within +/- 15mg/dL (<75mg/L YSI) or Within +/- 20% (>=75mg/dL YSI) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested Alternative Site (AST) palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS AST results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma BG results were used to calculate the number of AST BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma)
Time Frame: 1 hour
Population: 211 (219-8) Blood glucose results were analyzed. One subject discontinued from all testing after hypoglycemia Adverse Event. Three subjects with low blood sugar did not attempt palm testing per protocol. Two subjects had low blood sugar; their palm results were not evaluable per protocol. Two subjects failed to obtain palm blood for testing.
Measure: Number; unit: Blood Glucose results within 15mg/dL/20%
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 211
Blood Glucose results within 15mg/dL/20% | 209

5. Secondary Outcome: Number of Subject Fingerstick BG Results Within +/- 15mg/dL (<75mg/L YSI) or Within +/- 20% (>=75mg/dL YSI) of Laboratory Glucose Method When Tested by Study Staff
Description: Study staff tested subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results were used to calculate the number of BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) or +/- 20% (>=75mg/dL YSI capillary plasma)
Time Frame: 1 hour
Population: 218 (219-1) Blood glucose results were analyzed. One subject discontinued from testing after low BG result (hypoglycemia AE), thus no reference result available for that subject.
Measure: Number; unit: Blood Glucose results within 15mg/dL/20%
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 218
Blood Glucose results within 15mg/dL/20% | 218

6. Secondary Outcome: Number of Subject Responses That 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements
Description: Staff obtained subject responses using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' 'Agree' 'Neutral' 'Disagree' or 'Strongly Disagree'.
Time Frame: 1 hour
Population: 218 (219-1) responses were analyzed. One subject discontinued from testing after low BG result (hypoglycemia Adverse Event).
Measure: Number; unit: Participant Responses
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 218
Participant Responses
  I find it easy to do a blood test with this meter. | 218
  The meter display was easy to see and read. | 216
  It was easy to understand my test results. | 218
  I like the overall meter design. | 215
  I find the meter easy to use. | 217
  The instructions were easy to understand. | 213
  Instructions clearly explain how to run a test. | 216
  Instructions clearly explain meter error messages. | 217

ADVERSE EVENTS:
Time Frame: Subject visits were approximately 1 hour.
Arm/Group | Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/219
Other Adverse Events (participants affected / at risk) | 8/219
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Users of the Monitoring System (N=219)
Hypoglycemia (Endocrine disorders) | 8 (8) — Subjects' hypoglycemia events were resolved at the visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days